CLINICAL TRIAL: NCT01479491
Title: Observational Database Study on the Incidence of Intussusception in Children Aged < 12 Months in Japan
Brief Title: Study on the Incidence of Intussusception (IS) in Children Aged < 12 Months in Japan
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116259
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Intussusception
Keywords: Japan; Retrospective; Observational; Epidemiological study; Children aged < 12 months; Intussusception
MeSH Terms: conditions — Intussusception | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Case Group: Children aged < 12 months presenting with IS and covered by the Japan Medical Data Centre Company Limited (JMDC), Tokyo referred to as the JMDC Medical Data Bank (JMDC-MDB).
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data source will be the Japan Medical Data Centre Company Limited (JMDC) - JMDC Medical Data Bank (JMDC-MDB) database. Aggregated data (age in months and years and gender) for all subjects recorded in the database and subject-level data for IS cases will be extracted from the database. This database will be reviewed to extract data for the period between January 2005 and April 2011. Cases of IS will be identified using the International Classification of Diseases-10 (ICD-10) diagnostic codes, examination codes and procedural codes.

SUMMARY:
This study aims to analyse baseline data on IS in order to monitor the possibility of increased risk of IS in children aged <12 months after introduction of the Rotarix vaccination in Japan.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant aged < 12 months at the time of IS diagnosis and affiliated to the JMDC-MDB database.
* An IS case should be identified as per the ICD-10 diagnostic code-K56.1 (any-field listed), examination codes, and procedural codes.

Exclusion Criteria:

Not applicable

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged <12 months presenting with IS and covered by the JMDC-MDB database from January 2005 to April 2011.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of IS in subjects aged < 12 months | Between January 2005 and April 2011 (6 years)
Occurrence of age-specific and gender-specific incidence of IS among subjects aged < 12 months in Japan | Between January 2005 and April 2011 (6 years)

SECONDARY OUTCOMES:
Number of IS cases hospitalized more than once among subjects aged < 12 months. | Between January 2005 and April 2011 (6 years)
Occurrence of IS cases by calendar months and year among subjects aged < 12 months | Between January 2005 and April 2011 (6 years)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline